CLINICAL TRIAL: NCT04781413
Title: A Phase I/II, Single-center, Single-arm, Open-label Study of Nanoparticle Albumin-bound-paclitaxel (Nab-PTX) Plus S-1 and Sintilimab as Adjuvant Therapy in Patients With Stage IIIC Gastric Cancer
Brief Title: Nab-PTX Plus S-1 and Sintilimab as Adjuvant Therapy in Patients With Stage IIIC Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chair of Department of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON-VII
Record Dates: First submitted 2021-02-28; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Stage IIIC Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The phase I trial is a dose escalation design with standard 3+3 followed by expansion cohorts.
  Level Nab-PTX S-1 Sintilimab
  1. 80 mg/m2 80mg/m2 200mg
  2. 100 mg/m2 80mg/m2 200mg
  3. 120 mg/m2 80mg/m2 200mg
  We start at level 1. The recommended dose (RD) is defined as dose equal to the maximum tolerated dose (MTD). If 1 of three patients experiences dose-limiting toxicities (DLT), three more patients will be enrolled at the same dose level. The MTD is defined as the dose level at which two or more of three patients, or at least two of 4-6 patients, have DLTs during one cycle.
  Interventions: Drug: Nab-PTX, Sintilimab, S-1

INTERVENTIONS:
Drug: Nab-PTX, Sintilimab, S-1 — This is a single-arm study with all patients receiving these three drugs.

SUMMARY:
In this study, we combine Nab-PTX, S-1 and sintilimab as adjuvant regimen to patients with stage IIIC GC. We are aiming to investigate the recommended dose of this regimen in a phase I study and estimate the toxicity and efficacy of this regimen in a phase II study.

DETAILED DESCRIPTION:
The phase I study is a dose-escalation study using a standard 3+3 design. The regimen involves 3-week cycles with escalated doses of nab-paclitaxel (80-120 mg/m2 on days 1 and 8) and fixed doses of sintilimab (200 mg on day 1) and S-1 (based on body-surface area on day 1 to 14). The primary endpoints are safety and determination the recommended dose in the subsequent phase II study. In the phase II trial, the primary endpoint is 3-year relapse-free survival (RFS). Secondary endpoints are 5-year overall survival (OS), 3-year OS, 5-year RFS, and quality of life. Exploratory endpoint is time to peritoneal metastasis. Adverse events are monitored and graded according to the Common Terminology Criteria for Adverse Events version 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 80 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. Primary gastric cancer or gastroesophageal junction cancer that is pathologically diagnosed as adenocarcinoma;
4. Patients who have underwent radical resection with D2 lymphadenectomy and histologically proven to be stage IIIC gastric cancer according to the 8th edition of the UICC/AJCC TNM staging system for gastric cancer[29];
5. Patients who have received no prior chemotherapy or radiotherapy or immunotherapy for gastric cancer or gastroesophageal junction cancer;
6. No peritoneal metastasis by laparoscopy and no tumor cells in peritoneal fluid on cytologic analysis;
7. Adequate organ function for chemotherapy as follows:

   * absolute neutrophil count of ≥1.5×109/L;
   * platelet count of ≥100×109/L;
   * hemoglobin ≥90g/L;
   * bilirubin of <1.5×upper limit of normal [ULN];
   * alanine aminotransferase and aspartate aminotransferase of <2.5×ULN;
   * serum creatinine of ≤1.5×ULN;
   * creatinine clearance of >50 mL/min;
   * TSH ≤1×ULN (if abnormal, T3 and T4 levels should be inspected at the same time, if T3 and T4 levels are normal, they can be included in the group);
   * APTT ≤1.5×ULN and INR ≤1.5×ULN;
   * myocardial enzymogram ≤1×ULN.
8. Written (signed) informed consent;
9. Good compliance with the study procedures, including examination and treatment;
10. Surgeons should have experience doing this type of surgery (>50 procedures per year);
11. Patients have recovered from the operation and have no unresolved postoperative complications (such as postoperative infection, anastomotic leakage, gastrointestinal bleeding, pancreatic leakage) during baseline evaluation;
12. Start first treatment between 4 weeks and 12 weeks after surgery and there is no potential disease recurrence at the baseline evaluation;
13. The serum or urine HCG test of the female patients of non-surgical sterilization must be negative within 72 hours before the study group for the female patients of non-surgical sterilization or childbearing age;
14. During the study treatment period and within 3 months after the end of the study treatment period, a medically recognized contraceptive measure (such as IUD, contraceptive pill or condom) should be used for the enrolled patients.

Exclusion Criteria:

1. Distant metastatic disease evaluated by Chest-abdomen-pelvis CT, bone scan and head MR when with central nervous system symptoms or PET-CT;
2. R1 or R2 surgical margins;
3. Hospital stays exceeding 60 days;
4. Patients with history of prior or concurrent malignant tumors. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible;
5. Patients who received study drug treatment within 4 weeks before enrollment (participate in other clinical trials);
6. Patients with serious complications such as:

   * Uncontrolled cardiovascular disease, angina and arrhythmia;
   * Myocardial infarction in past six months;
   * Uncontrolled diabetes mellitus.
7. History of receiving anti-PD-1, anti-PD-L1, anti-PD-L2 or any other T cell co-simulation or checkpoint inhibitor therapy (eg. CTLA-4, OX-40, CD137);
8. Received any anti-cancer for this disease, including chemotherapy or radiotherapy or immunotherapy or Chinese traditional herb therapy;
9. Refuse to provide blood/tissue sample;
10. Female patients who are pregnant or lactating, or planning to become pregnant or lactating;
11. Active autoimmune disease or history of refractory autoimmune disease; Subjects with hypothyroidism requiring only hormone replacement therapy and skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia) can be selected;
12. Steroid or other systemic immunosuppressive therapy was used 14 days before admission, excluding local or physiological doses of systemic glucocorticoids (eg. no more than 10mg/day of prednisone or other glucocorticoids of equivalent dose) by nasal spray, inhalation or other routes, or hormones used to prevent allergy of contrast agents;
13. Uncontrollable pleural effusion, pericardial effusion or ascites;
14. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
15. Patients with history of hypersensitivity to any drugs in this study;
16. It may affect the absorption of S-1 in patients with upper gastrointestinal obstruction /bleeding, abnormal digestive function or malabsorption syndrome;
17. Have not fully recovered from toxicity or complications caused by any intervention before starting treatment;
18. HIV antibody positive, active hepatitis B or C (hepatitis B: HBsAg positive and HBV DNA ≥10 copies/ml; hepatitis C: HCV antibody and HCV-RNA positive, requiring antiviral treatment at the same time).
19. Receive live attenuated vaccine within 4 weeks before the first dose of study treatment or during the study period;
20. Severe or uncontrolled systemic disease:

    * severe cardiovascular diseases such as symptomatic coronary heart disease, congestive heart failure ≥ level II, uncontrolled arrhythmia and myocardial infarction within 12 months before admission;
    * active infection which requires systemic treatment;
    * active tuberculosis;
    * central nervous system (CNS) disorder or peripheral nervous system disorder or psychiatric disease;
    * history of primary immunodeficiency;
    * complicated with severe uncontrolled concurrent infection or other serious uncontrolled concomitant diseases, moderate or severe renal injury.
21. Other factors that may affect the safety or test compliance of the subjects according to the judgment of the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year relapse-free survival (RFS) | 36 months

SECONDARY OUTCOMES:
5-year overall survival (OS) | 60 months
5-year relapse-free survival (RFS) | 60 months
Adverse events | 36 months
  (based on Common Terminology Criteria for Adverse Events [CTCAE] version 4.0)
Peritoneal metastasis rate | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Zhu, Principal Investigator — Ruijin Hospital; Jun Zhang, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Surgery, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mei Y, Shi M, Zhu Z, Yuan H, Yan C, Li C, Feng T, Yan M, Zhang J, Zhu Z. Addition of sintilimab to nanoparticle albumin-bound paclitaxel and S-1 as adjuvant therapy in stage IIIC gastric cancer. Future Oncol. 2022 Jan;18(2):139-148. doi: 10.2217/fon-2021-1020. Epub 2021 Dec 8. PMID 34877867